CLINICAL TRIAL: NCT02406144
Title: Trial Studying Maintenance Treatment With Lenalidomide and Dexamethasone Versus Lenalidomide, Dexamethasone and MLN9708 After Autologous Hematopoietic Stem Cell Transplantation in Patients With Newly-diagnosed Symptomatic Multiple Myeloma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Celgene (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM2014MAIN
Record Dates: First submitted 2015-03-25; First posted 2015-04-02 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lenalidomide (Active Comparator): Oral administration of 15 mg/day of oral lenalidomide on days 1-21, and 20 mg/day of dexamethasone administered orally on days 1-4 and 9-12 for a period of two years
  Interventions: Drug: Lenalidomide; Drug: Dexamethasone
- MLN9708 plus Lenalidomide (Experimental): MLN9708 during the two year maintenance period, at a dose of 4 mg/day on days 1, 8 and 15 of the cycle.
  Interventions: Drug: MLN9708; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: MLN9708
  Arms: MLN9708 plus Lenalidomide
Drug: Lenalidomide
Drug: Dexamethasone

SUMMARY:
This protocol is a randomized, open-label, national, multicenter trial studying maintenance treatment with lenalidomide and dexamethasone versus lenalidomide, dexamethasone and MLN9708 after autologous hematopoietic stem cell transplantation in patients with newly-diagnosed symptomatic multiple myeloma.

A total of 316 patients, from the study GEM2012MENOS65, will be enrolled in the study.

The pre-treatment period includes the screening visit in which participants provide informed consent in writing in order to take part in the study. The patient is then assessed to determine his/her eligibility. The selection process will begin 21 days before the first dose of medication is administered (days -21 to 0). All procedures during the pre-treatment period will be carried out after completion of the two cycles of post-transplant consolidation with VRD which coincide with the end-of-study visit of clinical trial GEM2012MENOS65.

During the treatment period, eligible patients will be included in the study and receive maintenance treatment with lenalidomide/dexamethasone versus lenalidomide/dexamethasone/MLN9708. Each cycle will last 28 days. Treatment arm A will consist of oral administration of 15 mg/day of oral lenalidomide on days 1-21, and 20 mg/day of dexamethasone administered orally on days 1-4 and 9-12 for a period of two years. Arm B of the maintenance treatment will be the same as arm A, with the addition of MLN9708 during the two year maintenance period, at a dose of 4 mg/day on days 1, 8 and 15 of the cycle.

At two years, patients with negative MRD will finish maintenance treatment. Patients with positive MRD will continue treatment with lenalidomide/dexamethasone until they have completed five years of maintenance treatment. In this case, 20 mg/day of dexamethasone will only be administered on days 1-4 of the cycle. The dose of lenalidomide will not be adjusted. (unless necessary to treat adverse events)

Once this phase of active treatment is complete, patients will begin the long-term follow-up phase, during which they will be visited every three months to evaluate progression and survival.

DETAILED DESCRIPTION:
The primary trial objectives are:

• Impact on progression-free survival (PFS) when adding MLN9708 to post-transplant maintenance treatment with lenalidomide/dexamethasone in patients with multiple myeloma.

The secondary trial objectives are:

* Evaluate development and clinical significance of minimal residual disease (MRD) from the time maintenance treatment is initiated, yearly over five years.
* Overall survival (OS).
* Evaluate the safety and tolerability of the maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

* The patient must, in the opinion of the investigator, be capable of complying with all requirements of the trial.
* Have signed the informed consent form
* Be between 18 and 67 years of age
* Have an ECOG Performance Status <= 2 (or 3 if the ECOG is due to myeloma, e.g. pathological fracture)
* Multiple myeloma patient who was included in the GEM2012MENOS65 trial, and who is found to have, at a minimum, minimal response after consolidation
* Life expectancy > 3 months
* The patient must have the following laboratory values in the 21 days prior to initiation of treatment (day 1, cycle 1):

  1. Platelet count ≥ 100 x 109/L and absolute neutrophil count of ≥ 1.0 x 109/L. - Platelet transfusions to help patients meet eligibility criteria are not allowed.
  2. Corrected serum calcium < 14 mg/dL.
  3. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x the upper limit of normal (ULN)
  4. Total bilirubin within normal range
  5. Calculated creatinine clearance > 30 mL/min
* Female patients who:

  1. Are postmenopausal for at least 1 year before the screening visit, OR
  2. Are surgically sterile, OR
  3. If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 90 days after the last dose of study drug, AND
  4. Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR
  5. Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence [eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)
* Male patients, even if surgically sterilized (ie, status post-vasectomy), must agree to one of the following:

  1. Agree to practice effective barrier contraception during the entire study treatment period and through 90 days after the last dose of study drug, OR
  2. Must also adhere to the guidelines of any treatment-specific pregnancy prevention program, if applicable, OR 30 Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. (Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods] and withdrawal are not acceptable methods of contraception.)

Exclusion Criteria:

* Patients not included in clinical trial GEM2012MENOS65
* Patients included in GEM2012MENOS65 who are not found to have a least minimal response after consolidation
* Patients included in GEM2012MENOS65 who were discontinued prematurely due to toxicity or disease progression
* Female patients who are lactating or have a positive serum pregnancy test during the screening period.
* Central nervous system involvement
* Infection requiring systemic antibiotic therapy or other serious infection within 14 days before study enrollment.
* Systemic treatment, within 14 days before the first dose of MLN9708, with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin, ciprofloxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of MLN9708 including difficulty swallowing.
* Diagnosed or treated for another malignancy within 2 years before study enrollment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
* Peripheral neuropathy ≥ grade 2 in the 21 days prior to inclusion.
* Known hypersensitivity to lenalidomide or to MLN9708, their analogues, or excipients in the various formulations of any agent.
* Patients who have had a myocardial infarction in the six months prior to inclusion in the clinical trial, or who are class III or IV according to the New York Heart Association (NYHA), heart failure unstable angina, uncontrolled ventricular arrhythmias or acute ischemia detected by electrocardiogram, or conduction disorders.
* Patients who are currently participating in another clinical trial or receiving any other investigational product.
* Seropositive for HVB, HVC or HIV.

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 5 years
  Months to progression disease

SECONDARY OUTCOMES:
Minimal Residual Disease (MRD) | 5 years
  Number of patient with MRD and evaluation of its clinical significance
Overall survival | 6 years
  Months of survival

CONTACTS AND LOCATIONS:
Locations (74):
- Spain (74):
  - Complejo Hospitalario Universitario de Santiago, A Coruña
  - Hospital Txagorritxu, Alava
  - Hospital General de Albacete, Albacete
  - Hospital Del Vinalopo, Alicante
  - Hospital General Universitario de Alicante, Alicante
  - Hospital de Cabueñes, Asturias
  - Hospital Universitario Central de Asturias, Asturias
  - Hospital Clinic, Barcelona
  - H.Universitari Germans Trias I Pujol de Badalona, Barcelona
  - Hospital de La Santa Creu I Sant Pau, Barcelona
  - Hospital de Sabadell (Parc Taulí), Barcelona
  - Hospital de Sant Joan de Déu, Barcelona
  - Hospital Del Mar, Barcelona
  - Hospital Universitari Mútua de Terrasa, Barcelona
  - Hospital Vall D'Hebron, Barcelona
  - Ico L'Hospitalet, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital de Especialidades de Jerez de La Frontera, Cadiz
  - Hospital Universitario Marqués de Valdecilla, Cantabria
  - Hospital General de Castellón, Castelló
  - Complejo Hospitalario de Cáceres, Cáceres
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital Universitari Dr. Josep Trueta de Girona, Girona
  - Hospital de Gran Canaria Doctor Negrín, GRAN Canaria
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Universitario Guadalajara, Guadalajara
  - Hospital Universitario Donostia, Guipúzcoa
  - Hospital Son Llatzer, Illes Balears
  - Hospital Universitari Son Espases, Illes Balears
  - Hospital San Pedro, La Rioja
  - Hospital de León, León
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Centro Oncológico Md Anderson International España, Madrid
  - Fundación Jiménez Díaz-Ute, Madrid
  - Hm Universitario San Chinarro, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital de Fuenlabrada, Madrid
  - Hospital Del Tajo, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Infanta Sofía, Madrid
  - Hospital Ramón Y Cajal, Madrid
  - Hospital Severo Ochoa, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario Infanta Cristina, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Madrid
  - Complejo Hospital Costa Del Sol (Ivcs), Málaga
  - Hospital General Universitario Santa Lucia, Murcia
  - Hospital J.M. Morales Meseguer, Murcia
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Clinica Universidad de Navarra, Navarra
  - Complejo Hospitalario de Navarra, Navarra
  - Complejo Hospitalario de Ourense, Ourense
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital General de Segovia, Segovia
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Virgen del Rocío, Seville
  - Hospital Santa Bárbara, Soria
  - Hospital Universitari Joan Xxiii de Tarragona, Tarragona
  - Complejo Hospitalario de Toledo, Toledo
  - Hospital Nuestra Señora Del Prado, Toledo
  - Hospital Clínico Universitario Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario La Fe, Valencia
  - HOSPITAL CLíNICO UNIVERSITARIO DE VALLADOLID, Valladolid
  - Hospital Universitario Del Rio Hortega, Valladolid
  - Hospital de Cruces, Vizcaya
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Puig N, Agullo C, Contreras T, Cedena MT, Martinez-Lopez J, Oriol A, Blanchard MJ, Rios R, Inigo MB, Sureda A, Lakhwani S, de la Rubia J, Gonzalez-Calle V, Cabanas V, Palomera L, Moraleda JM, Bargay J, Castro S, Rosinol L, Blade J, San-Miguel JF, Lahuerta JJ, Paiva B, Mateos MV. Measurable residual disease by mass spectrometry and next-generation flow to assess treatment response in myeloma. Blood. 2024 Dec 5;144(23):2432-2438. doi: 10.1182/blood.2024024995. PMID 39293025
- [Derived] Guerrero C, Puig N, Cedena MT, Calasanz MJ, Gutierrez NC, Fernandez M, Oriol A, Rios-Tamayo R, Hernandez MT, Martinez-Martinez R, Bargay J, de Arriba F, Palomera L, Gonzalez-Rodriguez AP, Gonzalez Perez MS, Orfao A, Mateos MV, Martinez-Lopez J, Rosinol L, Blade J, Lahuerta JJ, San-Miguel JF, Paiva B. Predictors of unsustained measurable residual disease negativity in transplant-eligible patients with multiple myeloma. Blood. 2024 Feb 15;143(7):597-603. doi: 10.1182/blood.2023022083. PMID 38048552
- [Derived] Lakhwani S, Rosinol L, Puig N, Pico-Picos MA, Medina-Gonzalez L, Martinez-Lopez J, Paiva B, Cedena MT, Oriol A, Rios-Tamayo R, Blanchard MJ, Jarque I, Bargay J, Moraleda JM, Carrillo-Cruz E, Sureda A, Krsnik I, Gonzalez E, Casado LF, Marti JM, Encinas C, De Arriba F, Palomera L, Sampol A, Gonzalez-Montes Y, Motllo C, De La Cruz J, Alonso R, Mateos MV, Blade J, Lahuerta JJ, San-Miguel J, Hernandez MT. Recovery of uninvolved heavy/light chain pair immunoparesis in newly diagnosed transplant-eligible myeloma patients complements the prognostic value of minimal residual disease detection. Haematologica. 2024 Jun 1;109(6):1909-1917. doi: 10.3324/haematol.2023.284154. PMID 38031761
- [Derived] Rosinol L, Oriol A, Rios R, Blanchard MJ, Jarque I, Bargay J, Hernandez MT, Cabanas V, Carrillo-Cruz E, Sureda A, Martinez-Lopez J, Krsnik I, Gonzalez ME, Casado LF, Marti JM, Encinas C, de Arriba F, Palomera L, Sampol A, Gonzalez-Montes Y, Cabezudo E, Paiva B, Puig N, Cedena MT, de la Cruz J, Mateos MV, San Miguel J, Lahuerta JJ, Blade J. Lenalidomide and dexamethasone maintenance with or without ixazomib, tailored by residual disease status in myeloma. Blood. 2023 Nov 2;142(18):1518-1528. doi: 10.1182/blood.2022019531. PMID 37506339
- [Derived] Botta C, Maia C, Garces JJ, Termini R, Perez C, Manrique I, Burgos L, Zabaleta A, Alignani D, Sarvide S, Merino J, Puig N, Cedena MT, Rossi M, Tassone P, Gentile M, Correale P, Borrello I, Terpos E, Jelinek T, Paiva A, Roccaro A, Goldschmidt H, Avet-Loiseau H, Rosinol L, Mateos MV, Martinez-Lopez J, Lahuerta JJ, Blade J, San-Miguel JF, Paiva B. FlowCT for the analysis of large immunophenotypic data sets and biomarker discovery in cancer immunology. Blood Adv. 2022 Jan 25;6(2):690-703. doi: 10.1182/bloodadvances.2021005198. PMID 34587246